CLINICAL TRIAL: NCT04066933
Title: Neurogenic Thoracic Outlet Syndrome and Other Forms of Cervical Brachial Syndrome Treated With Plasma Concentrate Enriched for Alpha 2 Macroglobulin
Brief Title: Forms of Cervical Brachial Syndrome Treated With Plasma Concentrate Enriched for A2M
Acronym: A2M
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Neurological Associates of West Los Angeles (Other)
Responsible Party: Sponsor
Other Study IDs: 33237/1
Record Dates: First submitted 2019-08-19; First posted 2019-08-26 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Complex Regional Pain Syndromes; Neuralgia; Thoracic Outlet Neurologic Syndrome
Keywords: Alpha 2 macroglobulin
MeSH Terms: conditions — Complex Regional Pain Syndromes; Neuralgia; Thoracic Outlet Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: A2M enriched plasma — Plasma enriched for alpha2macroglobulin (A2M-PPP) was produced by a centrifugation and filtration process developed by Cytonics Corporation. Initially, 7 milliliters of Anticoagulant Citrate Dextrose Solution A, ubiquitous surface protein (USP) was drawn into a 60 cc syringe and then an additional 38 cc of autologous blood was drawn up through an antecubital vein. Two syringes were prepared in this manner and then centrifuged at 4000 rpm (1280G) for 4 minutes. The supernatant plasma fraction was then transferred to a roller pump system that circulates the fluid through a proprietary filter having a high molecular weight cutoff designed to trap larger molecules including alpha 2 macroglobulin (720 kDa).
  Other Names: A2M-PPP

SUMMARY:
Alpha 2 macroglobulin (A2M) is a plasma protein that acts as a molecular trap for inflammatory factors such as tumor necrosis factor (TNF). After plasma is enriched for A2M, it may be injected for treating chronic inflammation. Plasma enriched for A2M may be considered as a possible injectable agent to counteract inflammation that may occur with a cervicobrachial pain syndrome. This study reports on an experiencing using A2M to treat cervicobrachial syndrome which was predominant for either musculotendinous or neuralgic features.

DETAILED DESCRIPTION:
Regional pain in the neck, shoulder and arm is a common problem when there is exposure to repetitive work with a prevalence of about fifty percent. In the absence of a widespread pain conditions, and when cervical radiculopathy is ruled out with appropriate imaging, myalgia, tendinopathy or neurogenic sources of pain may predominate in a given case.

Myalgia (MTPS) may be characterized by muscles that are tight and tender to palpation and where there may be radiation of pain down the limb. A twitch may be elicited with stimulation of affected muscle. Numerous treatments for myalgia have been proposed with variable or incomplete success including local anesthetic injections, botulinum chemodenervation and platelet rich plasma injections.

Neuralgic complaints may be caused by chronic compression in the interscalene triangle as in Thoracic Outlet Syndrome (NTOS) and other patients may have injury from sudden stretch, electrocution, inflammatory diseases, penetrating wounds or acute or chronic post-operative conditions. Botulinum chemodenervation and surgical decompression has been applied for treating nerve compression due to Thoracic Outlet Syndrome with partial success. [9-13] Chemodenervation tends to be transient in effect and surgery may have significant complications.

Previous reports have demonstrated relatively poor outcomes with targeted treatments when there is a coexistence of conditions characterized by increased sensitivity as in complex regional pain syndrome (CRPS) or fibromyalgia. In the present retrospective review, it was anticipated that patients with CRPS may not respond as well to targeted treatment so that they were evaluated separately from patients with NTOS along.

Because existing therapies for myofascial and neuralgic forms of cervicobrachial pain may have unsatisfactory outcomes, alternative therapies may be considered, particularly, for individuals who have failed to respond. Contemporary conceptualizations of chronic pain mechanisms include the contribution of inflammatory factors. Mindful of these considerations, locally targeted anti-inflammatory administrations may be thought to play a potential role in treatment of cervicobrachial pain.

Alpha 2 macroglobulin is a plasma protein that acts as a molecular trap for inflammatory factors such as tumor necrosis factor, TNF. After plasma is enriched for A2M, it may be injected for treating chronic inflammation. Plasma enriched for A2M may be considered as a possible injectable agent to counteract inflammation that may occur with a cervicobrachial pain syndrome. The present paper reports on an experience using A2M for treating cervicobrachial syndrome which was predominant for either musculotendinous or neuralgic features.

ELIGIBILITY:
Inclusionary Criteria:

* All patients had daily disabling cervical brachial pain that was continuously present for at least six months.
* After examination by one or both of the authors, patients who were diagnosed as having a condition related to musculotendinous pain (MTPS), neuropathic Thoracic Outlet Syndrome (NTOS), or Complex Regional Pain Syndrome (CRPS) qualified for treatment and inclusion in the chart review.

Exclusionary Criteria:

* N/A
* (retrospective analysis of clinical treatment)

Ages: 23 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 56 patients (43 women, 13 men) with an age range of 23 to 77 years old who had undergone the outlined procedure were included in this chart review.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Brief Pain Inventory (BPI) | Baseline
  Self-report measure containing a composite pain score and functional interference score. The pain subscale contains 4 questions, each with answers ranging from 0 'no pain' to 10 'pain as bad as you can imagine.' Total possible score for the pain subscale is 40 points. The functional/interference subscale contains 7 questions, with each answer ranging from 0 'does not interfere' to 10 'completely interferes.' The maximum possible score for the interference subscale is 70 points. The total overall composite BPI score is out of 100 maximum points.
Patient Global Impression of Change Scale (PGIC) | 3 months
  Qualitative assessment of meaningful change obtained by a brief interview to estimate patients' overall perceived benefit of study procedures. The PGIC is structured as a 7-item scale ranging from 1 'very much improved' to 7 'very much worse.' Scores of 1 and 2 reflected notable subjective perception of benefit.

SECONDARY OUTCOMES:
Brief Pain Inventory (BPI) | 1 month
  Self-report measure containing a composite pain score and functional interference score. The pain subscale contains 4 questions, each with answers ranging from 0 'no pain' to 10 'pain as bad as you can imagine.' Total possible score for the pain subscale is 40 points. The functional/interference subscale contains 7 questions, with each answer ranging from 0 'does not interfere' to 10 'completely interferes.' The maximum possible score for the interference subscale is 70 points. The total overall composite BPI score is out of 100 maximum points. A clinical improvement is considered a decrease in BPI overall composite score by at least 30% from baseline.
Brief Pain Inventory (BPI) | 3 months
  Self-report measure containing a composite pain score and functional interference score. The pain subscale contains 4 questions, each with answers ranging from 0 'no pain' to 10 'pain as bad as you can imagine.' Total possible score for the pain subscale is 40 points. The functional/interference subscale contains 7 questions, with each answer ranging from 0 'does not interfere' to 10 'completely interferes.' The maximum possible score for the interference subscale is 70 points. The total overall composite BPI score is out of 100 maximum points. A clinical improvement is considered a decrease in BPI overall composite score by at least 30% from baseline.
Brief Pain Inventory (BPI) | 6 months
  Self-report measure containing a composite pain score and functional interference score. The pain subscale contains 4 questions, each with answers ranging from 0 'no pain' to 10 'pain as bad as you can imagine.' Total possible score for the pain subscale is 40 points. The functional/interference subscale contains 7 questions, with each answer ranging from 0 'does not interfere' to 10 'completely interferes.' The maximum possible score for the interference subscale is 70 points. The total overall composite BPI score is out of 100 maximum points. A clinical improvement is considered a decrease in BPI overall composite score by at least 30% from baseline.

OTHER OUTCOMES:
Adverse Event (AE) and Serious Adverse Event (SAE) Reporting | Reported throughout study duration, up to 12 months
  Any suspected adverse events possibly related to study procedures were noted. Any serious adverse events were reported immediately. [NONE REPORTED THROUGHOUT STUDY DURATION]

CONTACTS AND LOCATIONS:
Overall Officials: Sheldon Jordan, MD, FAAN, Principal Investigator — Neurological Associates of West Los Angeles
Locations (1):
- Neurological Associates of West Los Angeles, Santa Monica, California, United States

REFERENCES:
- [Background] Waersted M, Hanvold TN, Veiersted KB. Computer work and musculoskeletal disorders of the neck and upper extremity: a systematic review. BMC Musculoskelet Disord. 2010 Apr 29;11:79. doi: 10.1186/1471-2474-11-79. PMID 20429925
- [Background] Pascarelli EF, Hsu YP. Understanding work-related upper extremity disorders: clinical findings in 485 computer users, musicians, and others. J Occup Rehabil. 2001 Mar;11(1):1-21. doi: 10.1023/a:1016647923501. PMID 11706773
- [Background] Simons DG. The nature of myofascial trigger points. Clin J Pain. 1995 Mar;11(1):83-4. No abstract available. PMID 7787341
- [Background] Lavelle ED, Lavelle W, Smith HS. Myofascial trigger points. Med Clin North Am. 2007 Mar;91(2):229-39. doi: 10.1016/j.mcna.2006.12.004. PMID 17321283
- [Background] Cartagena-Sevilla J, Garcia-Fernandez MR, Vicente-Villena JP. Analgesic Effect of Botulinum Toxin A in Myofascial Pain Syndrome Patients Previously Treated with Local Infiltration of Anesthetic and Steroids. J Pain Palliat Care Pharmacother. 2016 Dec;30(4):269-275. doi: 10.1080/15360288.2016.1231742. Epub 2016 Nov 1. PMID 27802066
- [Background] Soares A, Andriolo RB, Atallah AN, da Silva EM. Botulinum toxin for myofascial pain syndromes in adults. Cochrane Database Syst Rev. 2014 Jul 25;2014(7):CD007533. doi: 10.1002/14651858.CD007533.pub3. PMID 25062018
- [Background] Tsikopoulos K, Tsikopoulos I, Simeonidis E, Papathanasiou E, Haidich AB, Anastasopoulos N, Natsis K. The clinical impact of platelet-rich plasma on tendinopathy compared to placebo or dry needling injections: A meta-analysis. Phys Ther Sport. 2016 Jan;17:87-94. doi: 10.1016/j.ptsp.2015.06.003. Epub 2015 Jun 18. PMID 26621224
- [Background] Jordan SE, Ahn SS, Gelabert HA. Combining ultrasonography and electromyography for botulinum chemodenervation treatment of thoracic outlet syndrome: comparison with fluoroscopy and electromyography guidance. Pain Physician. 2007 Jul;10(4):541-6. PMID 17660852
- [Background] Jordan SE, Ahn SS, Gelabert HA. Differentiation of thoracic outlet syndrome from treatment-resistant cervical brachial pain syndromes: development and utilization of a questionnaire, clinical examination and ultrasound evaluation. Pain Physician. 2007 May;10(3):441-52. PMID 17525778
- [Background] Christo PJ, Christo DK, Carinci AJ, Freischlag JA. Single CT-guided chemodenervation of the anterior scalene muscle with botulinum toxin for neurogenic thoracic outlet syndrome. Pain Med. 2010 Apr;11(4):504-11. doi: 10.1111/j.1526-4637.2010.00814.x. Epub 2010 Mar 1. PMID 20202146
- [Background] Torriani M, Gupta R, Donahue DM. Botulinum toxin injection in neurogenic thoracic outlet syndrome: results and experience using a ultrasound-guided approach. Skeletal Radiol. 2010 Oct;39(10):973-80. doi: 10.1007/s00256-010-0897-1. Epub 2010 Feb 26. PMID 20186413
- [Background] Thompson RW, Petrinec D. Surgical treatment of thoracic outlet compression syndromes: diagnostic considerations and transaxillary first rib resection. Ann Vasc Surg. 1997 May;11(3):315-23. doi: 10.1007/s100169900053. No abstract available. PMID 9140610
- [Background] Cuellar JM, Cuellar VG, Scuderi GJ. alpha2-Macroglobulin: Autologous Protease Inhibition Technology. Phys Med Rehabil Clin N Am. 2016 Nov;27(4):909-918. doi: 10.1016/j.pmr.2016.06.008. PMID 27788907
- [Background] Wang S, Wei X, Zhou J, Zhang J, Li K, Chen Q, Terek R, Fleming BC, Goldring MB, Ehrlich MG, Zhang G, Wei L. Identification of alpha2-macroglobulin as a master inhibitor of cartilage-degrading factors that attenuates the progression of posttraumatic osteoarthritis. Arthritis Rheumatol. 2014 Jul;66(7):1843-53. doi: 10.1002/art.38576. PMID 24578232
- [Background] Pasquale, X.M., Jason, M.C., Gaetano, J.S., Intradiscal injection of an Autologous Alpha-2-Macroglobulin (A2M) Concentrate Alleviates Back Pain in FAC-Positive Patients. Ortho and Rheum, 2017. 4(2).
- [Result] Eltayeb S, Staal JB, Kennes J, Lamberts PH, de Bie RA. Prevalence of complaints of arm, neck and shoulder among computer office workers and psychometric evaluation of a risk factor questionnaire. BMC Musculoskelet Disord. 2007 Jul 14;8:68. doi: 10.1186/1471-2474-8-68. PMID 17629925